CLINICAL TRIAL: NCT04833049
Title: A Phase 1 Study to Assess Absolute Bioavailability of TAK-994 and to Characterize Mass Balance, Pharmacokinetics, Absorption, Metabolism, and Excretion of [14C]TAK-994 in Male Healthy Subjects
Brief Title: Study to Evaluate Absorption, Metabolism, and Excretion, of TAK-994 in 6 Healthy Male Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: TAK-994-1004
Record Dates: First submitted 2021-04-05; First posted 2021-04-06 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAK-994 Dose 1 + [14C]TAK-994 Dose 2 + [14C]TAK-994 Dose 3 (Experimental): TAK-994 Dose 1, tablet, orally, on Day 1, followed by [14C]TAK-994 Dose 2, infusion, intravenously, on Day 1 of Part A, followed by a washout period of at least 8 days, further followed by [14C]TAK-994 Dose 3, suspension, orally, on Day 1 of Part B.
  Interventions: Drug: TAK-994 Oral Tablet; Drug: [14C]TAK-994 Intravenous Infusion; Drug: [14C]TAK-994 Oral Suspension

INTERVENTIONS:
Drug: TAK-994 Oral Tablet — TAK-994 tablet.
Drug: [14C]TAK-994 Intravenous Infusion — [14C]TAK-994 intravenous infusion.
Drug: [14C]TAK-994 Oral Suspension — [14C]TAK-994 oral suspension.

SUMMARY:
The aim of this study is to understand how TAK-994 is processed by the body.

This study will require participants to stay at the clinical research unit for 3 weeks to be monitored after receiving TAK-994.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-994. TAK-994 is being tested in healthy male participants. This study will characterize how TAK -994 is absorbed, metabolize, excreted by the body, after single oral administration by collecting plasma, urine, and feces samples for testing.

The study will enroll approximately 6 participants. The study consists of 2 parts: Part A and Part B.

In Part A, all participants will receive TAK-994 as tablet and [14C]TAK-994 as intravenous infusion. In Part B, all participants will receive a single dose of [14C]TAK-994 as an oral suspension.

This single-center trial will be conducted in the United States. The overall time to participate in this study is approximately 67 days, including a 28-day screening period plus approximately 30 days for follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) greater than or equal to (>=) 18.0 and less than (<) 32.0 kilogram per square meter (kg/m^2) at the screening.
2. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or electrocardiograms (ECGs), as deemed by the Investigator or designee.
3. Continuous non-smoker who has not used nicotine-containing products for at least 90 days prior to the first dosing and throughout the study, based on participant self-reporting.
4. Agrees to comply with any applicable contraceptive requirements of the protocol.
5. Agree not to donate sperm from the first dosing until 95 days after the last dosing.
6. Agree and able to remain in the clinical research unit (CRU) for the duration of the study.
7. Understands the study procedures in the ICF, and be willing and able to comply with the protocol.
8. Able to swallow oral suspensions.

Exclusion Criteria:

1. Mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the Investigator or designee.
3. History or presence of gastritis, gastrointestinal tract, hepatic disorder, cholecystectomy, history of treated or untreated Helicobacter pylori, ulcer disease, or other clinical condition which, in the opinion of the Investigator or designee, may affect the absorption, distribution, metabolism, or elimination of study drug.
4. History of any illness that, in the opinion of the Investigator or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
5. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing per the Diagnostic and Statistical Manual of Mental Disorders-V criteria.
6. History or presence of hypersensitivity or idiosyncratic reaction to the study drug or related compounds.
7. Current or past history of epilepsy, seizure, convulsion, tremor, or related symptoms.
8. Positive urine drug or alcohol results at screening or check-in.
9. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
10. Seated blood pressure is less than 90/40 millimeter of mercury (mmHg) or greater than 140/90 mmHg at screening.
11. Seated heart rate is lower than 45 beats per minute (bpm) or higher than 100 bpm at screening.
12. Orthostatic vital sign results with a decrease in systolic greater than (>) 20 mmHg or decrease in diastolic >10 mmHg, and increase in pulse of >20 bpm.
13. QT interval corrected for heart rate using Frederica's equation (QTcF) is >450 milliseconds (msec) or ECG findings are deemed abnormal with clinical significance by the Investigator or designee at screening.
14. Liver function tests including alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.5*upper limit of normal (ULN) at screening or check-in.
15. Estimated creatinine clearance <90 milliliter per minute (mL/min) at screening.
16. Tattoo(s) or scarring at or near the site of IV infusion or any other condition which may interfere with infusion site examination, in the opinion of the Investigator of designee;
17. Infrequent bowel movements (less than approximately once per day) within 30 days prior to dosing.
18. Recent history of abnormal bowel movements, such as diarrhea, loose stools, or constipation, within 2 weeks of dosing.
19. Lactose intolerance.
20. Has received radiolabeled substances or has been exposed to radiation sources within 12 months of first dosing or is likely to receive radiation exposure or radioisotopes within 12 months of last dosing such that participation in this study would increase their total exposure beyond the recommended levels considered safe (that is, weighted annual limit recommended by the International Commission on Radiological Protection [ICRP] of 3000 millirem [mrem]).
21. Unable to refrain from or anticipates the use of:

    * Any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements within 14 days prior to the first dosing and throughout the study. Thyroid hormone replacement medication may be permitted if the participant has been on the same stable dose for the immediate 3 months prior to first study drug administration. After first dosing and throughout the study, ibuprofen (up to 1.2 gram [g] per 24 hours) may be administered at the discretion of the Investigator or designee. Milk of Magnesia (that is, magnesium hydroxide) (less than or equal to [<=] 60 milliliter [mL] per day) may be administered from Day 3 of each study part, at discretion of the Investigator, to ensure defecation.
    * Any drugs known to be significant inducers or inhibitors of Cytochrome P450 3A4 (CYP3A4) enzymes and/or P-glycoprotein (P-gp), including St. John's Wort, within 28 days prior to the first dosing and throughout the study, including the follow-up period. Appropriate sources (example, Flockhart TableTM) will be consulted to confirm lack of pharmacokinetics (PK)/pharmacodynamics interaction with study drug.
22. Participation in another clinical study treated with the radiolabeled drug within 6 months prior to the first dosing.
23. Participants has a history of alcohol consumption exceeding 2 standard drinks per day on average (1 glass is approximately equivalent to the following: beer [354 mL/12 Ounce [oz]], wine [118 mL/4 oz], or distilled spirits [29.5 mL/1 oz] per day).
24. Participant consumes excessive amounts, defined as greater than 4 servings (1 serving is approximately equivalent to 120 mg of caffeine), of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.
25. Has been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to the first dosing and throughout the study.
26. Donation of blood or significant blood loss within 56 days prior to the first dosing.
27. Plasma donation within 7 days prior to the first dosing.
28. Participation in another clinical study within 30 days or 5 half-lives prior to the first dosing. The 30-day window or 5 half-lives will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Part A of the current study.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Part A: Percent Absolute Bioavailability (%F) for TAK-994 | Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
Part B: Percentage of Total Radioactivity (TRA) in Urine (Cum Percent [%] Dose [UR]) Relative to the Administered Radioactive Dose | Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Part B: Percentage of TRA in Feces (Cum%Dose[FE]) Relative to the Administered Radioactive Dose | Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Part B: Percentage of TRA Recovered in in the Urine and Feces Combined (Combined Cum%Dose) Relative to the Administered Radioactive Dose | Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose

SECONDARY OUTCOMES:
Part A, Ceoi: Plasma Concentration at the end of Infusion for [14C]TAK-994 | Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
Part A, CL: Total Clearance for [14C]TAK-994 | Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
Part A, Vss: Volume of Distribution at Steady State After Intravenous Administration for [14C]TAK-994 | Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
Part A, AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-994 and [14C]TAK-994 | Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
Part A, AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-994 and [14C]TAK-994 | Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
Part A, t(1/2z): Terminal Disposition Half-life for TAK-994 and [14C]TAK-994 | Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
Part A, Cmax: Maximum Observed Plasma Concentration for TAK-994 | Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
Part A, Tmax: Time to Reach the Maximum Plasma Concentration for TAK-994 | Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
Part B, Cmax: Maximum Observed Plasma Concentration for TAK-994 | Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Part B, Tmax: Time to Reach the Maximum Plasma Concentration for TAK-994 | Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Part B, AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-994 | Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Part B, AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-994 | Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Part B, t(1/2z): Terminal Disposition Half-life for TAK-994 | Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Part B, Cmax: Maximum Observed Plasma and Whole Blood TRA Concentration for TAK-994 | Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Part B, Tmax: Time to Reach the Maximum Plasma and Whole Blood TRA Concentration (Cmax) for TAK-994 | Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Part B, AUClast: Area Under the Plasma and Whole Blood TRA Concentration-time Curve From Time 0 to Last Quantifiable Concentration for TAK-994 | Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Part B, AUC∞: Area Under the Plasma and Whole Blood TRA Concentration-time Curve From Time 0 to Infinity for TAK-994 | Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Part B, AUCt: Area Under the Plasma and Whole Blood TRA Concentration-time Curve From Time 0 to Time t for TAK-994 | Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Part B, t(1/2z): Terminal Disposition Phase Half-life of Plasma and Whole Blood TRA Concentration for TAK-994 | Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/606d6838620b3b001e9dbb5c